CLINICAL TRIAL: NCT07271277
Title: 3D MRI Assessment of Femoroacetabular Impingement in Patients With ACL Rupture - Exploratory Study
Acronym: IMAHANCHE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-A01269-40
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Femoroacetabular Impingement
Keywords: femoroacetabular impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAI arm (Experimental): FAI arm involves patients with ACL rupture. A 3D MRI scan of both hips of theses patients will be performed.
  Interventions: Other: 3D MRI

INTERVENTIONS:
Other: 3D MRI — Intervention consists of performing a 3D MRI scan of both hips using a T1 sequence.

SUMMARY:
Anterior cruciate ligament (ACL) tears are among the most common sports injuries. Numerous studies have shown that reduced hip rotation may play a role in ACL tears. The same question may also arise for hip injuries such as femoroacetabular impingement (FAI).

This research is based on the hypothesis that there is a relationship between FAI and ACL injury. In this context, 3D MRI of the hip would provide morphological details of the hip that are not currently available with other imaging techniques, thereby enabling early identification of FAI. This is the reason why this research has been initiated.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) tears are among the most common sports injuries. It is estimated that approximately 150,000 ACL reconstructions are performed each year in the United States. Numerous studies have shown that reduced hip rotation may play a role in ACL tears. The same question may also arise for hip injuries such as femoroacetabular impingement (FAI).

This research is based on the hypothesis that there is a relationship between FAI and ACL injury. In this context, 3D MRI of the hip would provide morphological details of the hip that are not currently available with other imaging techniques, thereby enabling early identification of FAI. This is the reason why this research has been initiated.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged 18 years or older
* Patient with a primary complete ACL rupture
* Patient affiliated with or covered by a social security scheme
* Patient who speaks French and has signed an informed consent form

Exclusion Criteria:

* Patient with multi-ligament injury
* Patients with a history of hip fracture
* Patients with a history of hip surgery
* Patients with a contraindication to MRI
* Protected individuals: adults under guardianship, curatorship or other legal protection, deprived of their liberty by judicial or administrative decision
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
FAI (femoroacetabular impingement) prevalence | Day 1
  Prevalence of femoroacetabular impingement will be expressed as %. It will be measured on the injured knee side (i.e., ACL rupture) and on the healthy knee side (i.e., uninjured).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, France, France

IPD SHARING:
Plan to Share IPD: No